CLINICAL TRIAL: NCT04337853
Title: Implementation of an Intraoral Stent in Radiotherapy of Tongue Cancer
Brief Title: Radiotherapy of Tongue Cancer Using an Intraoral Stent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Einar Dale, Senior Consultant, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-139
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Tongue Cancer
Keywords: Radiotherapy; Head and neck cancer; Intraoral stent
MeSH Terms: conditions — Tongue Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): N=6
  Interventions: Device: Intraoral stent
- Control group (Active Comparator): N=7
  Interventions: Other: No intraoral stent

INTERVENTIONS:
Device: Intraoral stent — Radiotherapy with intraoral stent
  Arms: Intervention group
Other: No intraoral stent — Radiotherapy without intraoral stent
  Arms: Control group

SUMMARY:
Radiotherapy of tongue cancer is associated with acute and late morbidity. Use of an intraoral stent will provide a larger distance between the tongue and palate and can reduce side-effects. The aim of the present study is to confirm that an intraoral stent will give lower dose to the palate throughout the treatment period.

DETAILED DESCRIPTION:
Radiotherapy of tongue cancer is associated with acute and late morbidity. Use of an intraoral stent will provide a larger distance between the tongue and palate and can reduce side-effects. The main objective of the present study is to confirm that the use of an intraoral stent will result in lower dose to the palate throughout the treatment period. A secondary objective is to measure the reduction in acute mucositis in the palate.

The intraoral stent used in the present study is available in two sizes, 10 and 20mm thickness. The intervention group and control group will consist of approximately five patients each. Target coverage will be measured by the minimum dose covering 98% of the clinical target volume (D98CTV). Dose to the organs at risk (hard and soft palate) will be measured by the mean dose. Data will be collected from the planning computed tomography (CT) and daily cone-beam CT (CBCT). Acute mucositis will be scored by Common Terminology Criteria for Adverse Events (CTCAE) v3.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tongue cancer
* Curatively intended radiotherapy requiring a total dose of 50-70 Gy
* Age >18 years
* Performance status, Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Reduction in mean dose to the hard palate | At the end of radiotherapy (5-6 weeks)
  Mann-Whitney U test.

SECONDARY OUTCOMES:
Reduction in mean dose to the soft palate | At the end of radiotherapy (5-6 weeks)
  Mann-Whitney U test.
Reduction in acute mucositis in the hard palate | At the end of radiotherapy (5-6 weeks)
  CTCAE score in the hard palate. Mann-Whitney U test.
Reduction in acute mucositis in the soft palate | At the end of radiotherapy (5-6 weeks)
  CTCAE score in the hard palate. Mann-Whitney U test.

CONTACTS AND LOCATIONS:
Overall Officials: Einar Dale, MD PhD, Principal Investigator — Oslo University Hospital, Department of Oncology
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results — https://www.cambridge.org/core/journals/journal-of-radiotherapy-in-practice/article/radiotherapy-of-tongue-cancer-using-an-intraoral-stent-a-pilot-study/EA0903883867854A0190757E4CF9777A